CLINICAL TRIAL: NCT02467179
Title: Evaluation of the Amigo Robotic System for Ablation of the Cavo-Tricuspid Isthmus
Acronym: Amigo-AFL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Catheter Robotics, Inc. (Industry)
Responsible Party: Principal Investigator, Gregory Kent Feld, Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 150318
Record Dates: First submitted 2015-06-03; First posted 2015-06-09 (Estimated); Results first posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: Arrhythmia; cavo-tricuspid isthmus; atrial fibrillation; atrial fibrillation ablation
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Arrhythmias, Cardiac | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual Catheter Manipulation (Active Comparator): 25 subjects will be randomized to this arm. Manual catheter ablation of the cavo-tricuspid isthmus will be performed.
  Interventions: Device: Manual Catheter Manipulation
- Amigo™ Robotic Catheter Manipulation (Experimental): 25 subjects will be randomized to this arm. Robotic catheter ablation of the cavo-tricuspid isthmus with the Amigo Catheter System will be performed.
  Interventions: Device: Amigo™ Robotic Catheter Manipulation

INTERVENTIONS:
Device: Amigo™ Robotic Catheter Manipulation — Ablation is a standard procedure that patients may undergo for the atrial flutter.
  In this study, this group will be assigned to robotic catheter manipulation.
  Other Names: cavo-tricuspid isthmus ablation; atrial flutter ablation; arrhythmia; radiofrequency catheter ablation
  Arms: Amigo™ Robotic Catheter Manipulation
Device: Manual Catheter Manipulation — Ablation is a standard procedure that patients may undergo for the atrial flutter.
  In this study, this group will be assigned to manual catheter manipulation.
  Other Names: cavo-tricuspid isthmus ablation; atrial flutter ablation; arrhythmia; radiofrequency catheter ablation
  Arms: Manual Catheter Manipulation

SUMMARY:
The purpose of this study is to compare standard manual and robotically controlled catheter ablation of the cavo-tricuspid isthmus (CTI) as a treatment for atrial flutter. Ablation of the CTI is standard treatment for patients with a history of atrial flutter, and those undergoing ablation for atrial fibrillation. Both manual and robotic catheter manipulation are used in standard clinical practice at The University of California, San Diego (UCSD) for ablation.

DETAILED DESCRIPTION:
Dr. Gregory Feld, M.D. is conducting a research study to find out more about the effects of using the Amigo™ Robotic System for ablation of the cavo-tricuspid isthmus (flutter isthmus) on catheter stability (stabilization of the catheter during the procedure in order to prevent movement and dislodgement) using a combination of contact force (a measurement of the force applied by the catheter tip against the tissue during the ablation procedure), location, and duration measurements during ablation of the atrial flutter circuit. Published studies have indicated that robotic catheter manipulation is safe, may reduce patient and physician x-ray exposure, and ablation procedure time. Measuring contact force has also been shown to improve both short-term and long-term procedure success. However, research on ablation of the CTI specifically, is limited. This is a randomized study comparing robotic catheter manipulation using the Amigo Robotic System to manual catheter manipulation for ablation of the CTI on measures including catheter stability, contact force, procedure time, and fluoroscopy (X-ray) time.

The ablation procedure is standard of care, however, if patients chose to enroll in the study they will be randomized to one of two groups: either manual or robotic catheter manipulation. Throughout the procedure, research personnel will collect information from the procedure including measurements of contact force, catheter stability, procedure duration, and fluoroscopy (X-ray) time. If, in addition to ablation of the cavo-tricuspid isthmus for atrial flutter, a patient is scheduled to undergo ablation of the left atrium for atrial fibrillation or left atrial flutter, this will be performed subsequently in a standard manner, and will not be considered part of the research. Ablation of the CTI generally takes 45-60 minutes regardless of the technique used for manipulation of the catheters.

The patient's participation in the study will only last one day, the length of study procedure. There is no follow up associated with this study. All subjects will received standard of care treatment following their ablation.

ELIGIBILITY:
Inclusion Criteria:

* Must be scheduled to undergo radiofrequency catheter ablation of the cavo-tricuspid isthmus for atrial fibrillation (AF) or atrial flutter (AFL) according to appropriate clinical indications.
* Must be able and willing to provide written informed consent
* Must be at least 18 years old.

Exclusion Criteria:

* Patient's refusal to participate in the study
* Lack of indication for CTI ablation (eg: prior CTI ablation with persistent bidirectional isthmus block)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Feld, MD, Principal Investigator — UC San Diego
Locations (1):
- Sulpizio Cardiovascular Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wood MA, Orlov M, Ramaswamy K, Haffajee C, Ellenbogen K; Stereotaxis Heart Study Investigators. Remote magnetic versus manual catheter navigation for ablation of supraventricular tachycardias: a randomized, multicenter trial. Pacing Clin Electrophysiol. 2008 Oct;31(10):1313-21. doi: 10.1111/j.1540-8159.2008.01183.x. PMID 18811813
- [Result] Proietti R, Pecoraro V, Di Biase L, Natale A, Santangeli P, Viecca M, Sagone A, Galli A, Moja L, Tagliabue L. Remote magnetic with open-irrigated catheter vs. manual navigation for ablation of atrial fibrillation: a systematic review and meta-analysis. Europace. 2013 Sep;15(9):1241-8. doi: 10.1093/europace/eut058. Epub 2013 Apr 12. PMID 23585253
- [Result] Hlivak P, Mlcochova H, Peichl P, Cihak R, Wichterle D, Kautzner J. Robotic navigation in catheter ablation for paroxysmal atrial fibrillation: midterm efficacy and predictors of postablation arrhythmia recurrences. J Cardiovasc Electrophysiol. 2011 May;22(5):534-40. doi: 10.1111/j.1540-8167.2010.01942.x. Epub 2010 Nov 23. PMID 21091964
- [Result] Feld G, Wharton M, Plumb V, Daoud E, Friehling T, Epstein L; EPT-1000 XP Cardiac Ablation System Investigators. Radiofrequency catheter ablation of type 1 atrial flutter using large-tip 8- or 10-mm electrode catheters and a high-output radiofrequency energy generator: results of a multicenter safety and efficacy study. J Am Coll Cardiol. 2004 Apr 21;43(8):1466-72. doi: 10.1016/j.jacc.2003.11.036. PMID 15093885
- [Result] Sawhney N, Anousheh R, Chen WC, Narayan S, Feld GK. Five-year outcomes after segmental pulmonary vein isolation for paroxysmal atrial fibrillation. Am J Cardiol. 2009 Aug 1;104(3):366-72. doi: 10.1016/j.amjcard.2009.03.044. Epub 2009 Jun 6. PMID 19616669
- [Result] Steinberg JS, Palekar R, Sichrovsky T, Arshad A, Preminger M, Musat D, Shaw RE, Mittal S. Very long-term outcome after initially successful catheter ablation of atrial fibrillation. Heart Rhythm. 2014 May;11(5):771-6. doi: 10.1016/j.hrthm.2014.02.003. Epub 2014 Feb 4. PMID 24508206
- [Result] Akca F, Janse P, Theuns DA, Szili-Torok T. A prospective study on safety of catheter ablation procedures: contact force guided ablation could reduce the risk of cardiac perforation. Int J Cardiol. 2015 Jan 20;179:441-8. doi: 10.1016/j.ijcard.2014.11.105. Epub 2014 Nov 13. PMID 25465303
- [Result] Sigmund E, Puererfellner H, Derndorfer M, Kollias G, Winter S, Aichinger J, Nesser HJ, Martinek M. Optimizing radiofrequency ablation of paroxysmal and persistent atrial fibrillation by direct catheter force measurement-a case-matched comparison in 198 patients. Pacing Clin Electrophysiol. 2015 Feb;38(2):201-8. doi: 10.1111/pace.12549. Epub 2014 Dec 2. PMID 25469738
- [Result] Jarman JWE, Panikker S, DAS M, Wynn GJ, Ullah W, Kontogeorgis A, Haldar SK, Patel PJ, Hussain W, Markides V, Gupta D, Schilling RJ, Wong T. Relationship between contact force sensing technology and medium-term outcome of atrial fibrillation ablation: a multicenter study of 600 patients. J Cardiovasc Electrophysiol. 2015 Apr;26(4):378-384. doi: 10.1111/jce.12606. Epub 2015 Feb 11. PMID 25546580
- [Result] le Polain de Waroux JB, Weerasooriya R, Anvardeen K, Barbraud C, Marchandise S, De Meester C, Goesaert C, Reis I, Scavee C. Low contact force and force-time integral predict early recovery and dormant conduction revealed by adenosine after pulmonary vein isolation. Europace. 2015 Jun;17(6):877-83. doi: 10.1093/europace/euu329. Epub 2015 Jan 24. PMID 25618742
- [Result] Arujuna A, Karim R, Zarinabad N, Gill J, Rhode K, Schaeffter T, Wright M, Rinaldi CA, Cooklin M, Razavi R, O'Neill MD, Gill JS. A randomized prospective mechanistic cardiac magnetic resonance study correlating catheter stability, late gadolinium enhancement and 3 year clinical outcomes in robotically assisted vs. standard catheter ablation. Europace. 2015 Aug;17(8):1241-50. doi: 10.1093/europace/euu364. Epub 2015 Feb 16. PMID 25687748
- [Result] Shurrab M, Danon A, Lashevsky I, Kiss A, Newman D, Szili-Torok T, Crystal E. Robotically assisted ablation of atrial fibrillation: a systematic review and meta-analysis. Int J Cardiol. 2013 Nov 5;169(3):157-65. doi: 10.1016/j.ijcard.2013.08.086. Epub 2013 Sep 10. PMID 24063921
- [Result] Lopez-Gil M, Salgado R, Merino JL, Datino T, Figueroa J, Arenal A, Mejia E, Salguero R, Fontenla A, Arribas F. Cavo-tricuspid isthmus radiofrequency ablation using a novel remote navigation catheter system in patients with typical atrial flutter. Europace. 2014 Apr;16(4):558-62. doi: 10.1093/europace/eut285. Epub 2013 Sep 20. PMID 24058180
- [Result] Datino T, Arenal A, Pelliza M, Hernandez-Hernandez J, Atienza F, Gonzalez-Torrecilla E, Avila P, Bravo L, Fernandez-Aviles F. Comparison of the safety and feasibility of arrhythmia ablation using the Amigo Robotic Remote Catheter System versus manual ablation. Am J Cardiol. 2014 Mar 1;113(5):827-31. doi: 10.1016/j.amjcard.2013.11.030. Epub 2013 Dec 12. PMID 24440330
- [Result] Zhang W, Jia N, Su J, Lin J, Peng F, Niu W. The comparison between robotic and manual ablations in the treatment of atrial fibrillation: a systematic review and meta-analysis. PLoS One. 2014 May 6;9(5):e96331. doi: 10.1371/journal.pone.0096331. eCollection 2014. PMID 24800808
- [Result] Wutzler A, Wolber T, Parwani AS, Huemer M, Attanasio P, Blaschke F, Haegeli L, Haverkamp W, Duru F, Boldt LH. Robotic ablation of atrial fibrillation with a new remote catheter system. J Interv Card Electrophysiol. 2014 Sep;40(3):215-9. doi: 10.1007/s10840-014-9895-x. Epub 2014 Apr 29. PMID 24771262
- [Result] Thomas D, Scholz EP, Schweizer PA, Katus HA, Becker R. Initial experience with robotic navigation for catheter ablation of paroxysmal and persistent atrial fibrillation. J Electrocardiol. 2012 Mar;45(2):95-101. doi: 10.1016/j.jelectrocard.2011.05.005. Epub 2011 Jun 28. PMID 21714971
- [Derived] Hoffmayer KS, Krainski F, Shah S, Hunter J, Alegre M, Hsu JC, Feld GK. Randomized controlled trial of Amigo(R) robotically controlled versus manually controlled ablation of the cavo-tricuspid isthmus using a contact force ablation catheter. J Interv Card Electrophysiol. 2018 Mar;51(2):125-132. doi: 10.1007/s10840-018-0319-1. Epub 2018 Feb 12. PMID 29435790

RESULTS

PARTICIPANT FLOW:
Groups:
- Manual Catheter Manipulation: 25 subjects will be randomized to this arm. Manual catheter ablation of the cavo-tricuspid isthmus will be performed.
  Manual Catheter Manipulation: Ablation is a standard procedure that patients may undergo for the atrial flutter.
  In this study, this group will be assigned to manual catheter manipulation.
- Amigo™ Robotic Catheter Manipulation: 25 subjects will be randomized to this arm. Robotic catheter ablation of the cavo-tricuspid isthmus with the Amigo Catheter System will be performed.
  Amigo™ Robotic Catheter Manipulation: Ablation is a standard procedure that patients may undergo for the atrial flutter.
  In this study, this group will be assigned to robotic catheter manipulation.
Period: Overall Study
Arm/Group | Manual Catheter Manipulation | Amigo™ Robotic Catheter Manipulation
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Manual Catheter Manipulation | Amigo™ Robotic Catheter Manipulation | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (12) | 63 (12) | 63 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 17 | 19 | 36
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Contact Force Through Measurement of Force-time Integral (FTI)
Description: Determination of the average total contact force (measured in gs) achieved during each ablation lesion using the Carto Mapping System
Time Frame: At time of the ablation procedure, which typically lasts 30-60 minutes
Measure: Mean (Standard Deviation); unit: gm/s
Arm/Group | Manual Catheter Manipulation | Amigo™ Robotic Catheter Manipulation
Number analyzed (Participants) | 25 | 25
gm/s | 471 (179) | 571 (278)

2. Secondary Outcome: Fluoroscopy Time Measurements
Description: Determine fluoroscopy time to reach CTI block.
Time Frame: at time of ablation procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Manual Catheter Manipulation | Amigo™ Robotic Catheter Manipulation
Number analyzed (Participants) | 25 | 25
minutes | 3.8 (2.3) | 6.8 (4.4)

ADVERSE EVENTS:
Time Frame: From the time of enrollment to completion of the ablation procedure (which usually lasted 30-60 minutes).
Arm/Group | Manual Catheter Manipulation | Amigo™ Robotic Catheter Manipulation
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2015-03-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT02467179/Prot_000.pdf